CLINICAL TRIAL: NCT01736449
Title: Role of Sub-Conjunctival Bevacizumab in Post Pterygium Excision Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Principal Investigator, Sonia Dhoot, Prinicipal Investigator, Arrowhead Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB1108
Record Dates: First submitted 2012-11-21; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Pterygium
Keywords: pterygium; bevacizumab; recurrence of pterygium
MeSH Terms: conditions — Pterygium | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pterygium Excision Alone (Placebo Comparator)
- Pterygium Excision with Bevacizumab Injection (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
  Arms: Pterygium Excision with Bevacizumab Injection

SUMMARY:
A pterygium is a fibrovascular growth originating from the conjunctiva that grows onto the surface of the cornea. Frequently, these pterygia will recur even after surgical resection. Bevacizumab is an inhibitor of angiogenesis, which is needed for recurrent growth. The use of bevacizumab is poorly understood in inhibiting pterygium growth. The objective of this study is to compare the effects of wound healing and recurrence rates in postoperative bevacizumab versus pterygium excision alone.

DETAILED DESCRIPTION:
This is a prospective trial. Thirty-one patients with a primary pterygium of at least 2 mm in size and without any previous ocular surgery will be included. Outcome measures will include best corrected visual acuity, intraocular pressure, recurrence, and any sight threatening complications at two weeks, two months, and six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* any patient 18 years of age or older with a primary pterygium that extends at least 2 mm past the limbus

Exclusion Criteria:

* history of glaucoma
* previous ocular surgery
* steroid-response glaucoma
* previous myocardial infarct
* bleeding disorder
* pregnancy
* lack of patient cooperation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
number of recurrent pterygia with postoperative bevacizumab | 6 months
  The number of recurrent pterygia with patients who received bevacizumab after pterygium excision was compared to the number of recurrences in those patients who only had pterygium excision.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Tokuhara, MD, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

REFERENCES:
- [Background] Detorakis ET, Spandidos DA. Pathogenetic mechanisms and treatment options for ophthalmic pterygium: trends and perspectives (Review). Int J Mol Med. 2009 Apr;23(4):439-47. doi: 10.3892/ijmm_00000149. PMID 19288018
- [Background] Detorakis ET, Zaravinos A, Spandidos DA. Growth factor expression in ophthalmic pterygia and normal conjunctiva. Int J Mol Med. 2010 Apr;25(4):513-6. doi: 10.3892/ijmm_00000371. PMID 20198298
- [Background] Avisar R, Arnon A, Avisar E, Weinberger D. Primary pterygium recurrence time. Isr Med Assoc J. 2001 Nov;3(11):836-7. PMID 11729580
- [Background] Hirst LW. The treatment of pterygium. Surv Ophthalmol. 2003 Mar-Apr;48(2):145-80. doi: 10.1016/s0039-6257(02)00463-0. PMID 12686302
- [Background] Ang LP, Chua JL, Tan DT. Current concepts and techniques in pterygium treatment. Curr Opin Ophthalmol. 2007 Jul;18(4):308-13. doi: 10.1097/ICU.0b013e3281a7ecbb. PMID 17568207
- [Background] Enkvetchakul O, Thanathanee O, Rangsin R, Lekhanont K, Suwan-Apichon O. A randomized controlled trial of intralesional bevacizumab injection on primary pterygium: preliminary results. Cornea. 2011 Nov;30(11):1213-8. doi: 10.1097/ICO.0b013e31821c9b44. PMID 21915047
- [Background] Fallah Tafti MR, Khosravifard K, Mohammadpour M, Hashemian MN, Kiarudi MY. Efficacy of intralesional bevacizumab injection in decreasing pterygium size. Cornea. 2011 Feb;30(2):127-9. doi: 10.1097/ICO.0b013e3181e16d67. PMID 20885313
- [Background] Banifatemi M, Razeghinejad MR, Hosseini H, Gholampour A. Bevacizumab and ocular wound healing after primary pterygium excision. J Ocul Pharmacol Ther. 2011 Feb;27(1):17-21. doi: 10.1089/jop.2010.0094. Epub 2010 Oct 26. PMID 20977367
- [Background] Razeghinejad MR, Hosseini H, Ahmadi F, Rahat F, Eghbal H. Preliminary results of subconjunctival bevacizumab in primary pterygium excision. Ophthalmic Res. 2010;43(3):134-8. doi: 10.1159/000252980. Epub 2009 Oct 29. PMID 19887878
- [Background] Lekhanont K, Patarakittam T, Thongphiew P, Suwan-apichon O, Hanutsaha P. Randomized controlled trial of subconjunctival bevacizumab injection in impending recurrent pterygium: a pilot study. Cornea. 2012 Feb;31(2):155-61. doi: 10.1097/ICO.0b013e3182151e0e. PMID 22081150
- [Background] Fallah MR, Khosravi K, Hashemian MN, Beheshtnezhad AH, Rajabi MT, Gohari M. Efficacy of topical bevacizumab for inhibiting growth of impending recurrent pterygium. Curr Eye Res. 2010 Jan;35(1):17-22. doi: 10.3109/02713680903395273. PMID 20021250
- [Background] Shenasi A, Mousavi F, Shoa-Ahari S, Rahimi-Ardabili B, Fouladi RF. Subconjunctival bevacizumab immediately after excision of primary pterygium: the first clinical trial. Cornea. 2011 Nov;30(11):1219-22. doi: 10.1097/ICO.0b013e31820ca63f. PMID 21955635
- [Background] Cortez RT, Ramirez G, Collet L, Thakuria P, Giuliari GP. Intravitreous bevacizumab injection: an experimental study in New Zealand white rabbits. Arch Ophthalmol. 2010 Jul;128(7):884-7. doi: 10.1001/archophthalmol.2010.139. PMID 20625050
- [Background] Michels S. Is intravitreal bevacizumab (Avastin) safe? Br J Ophthalmol. 2006 Nov;90(11):1333-4. doi: 10.1136/bjo.2006.102293. PMID 17057166
- [Background] Ghazi NG, Kirk TQ, Knape RM, Tiedeman JS, Conway BP. Is monthly retreatment with intravitreal bevacizumab (Avastin) necessary in neovascular age-related macular degeneration? Clin Ophthalmol. 2010 Apr 26;4:307-14. doi: 10.2147/opth.s8598. PMID 20463798
- [Background] El-Batarny AM. Intravitreal bevacizumab treatment for retinal neovascularization and vitreous hemorrhage in proliferative diabetic retinopathy. Clin Ophthalmol. 2007 Jun;1(2):149-55. PMID 19668504
- [Background] Wong D, Joussen AM. The safety of using anti-VEGF: Is there strength in numbers? Curtis LH, Hammill BG, Schulman KA, Cousins SW (2010) Risks of mortality, myocardial infarction, bleeding, and stroke associated with therapies for age-related macular degeneration. Arch Ophthalmol 128(10):1273-1279. Graefes Arch Clin Exp Ophthalmol. 2011 Feb;249(2):161-2. doi: 10.1007/s00417-010-1603-7. Epub 2011 Jan 6. No abstract available. PMID 21210141
- [Background] Grisanti S, Ziemssen F. Bevacizumab: off-label use in ophthalmology. Indian J Ophthalmol. 2007 Nov-Dec;55(6):417-20. doi: 10.4103/0301-4738.36474. PMID 17951896
- [Background] Yazdani S, Hendi K, Pakravan M. Intravitreal bevacizumab (Avastin) injection for neovascular glaucoma. J Glaucoma. 2007 Aug;16(5):437-9. doi: 10.1097/IJG.0b013e3180457c47. PMID 17700285
- [Background] Arevalo JF, Sanchez JG, Lasave AF, Wu L, Maia M, Bonafonte S, Brito M, Alezzandrini AA, Restrepo N, Berrocal MH, Saravia M, Farah ME, Fromow-Guerra J, Morales-Canton V. Intravitreal Bevacizumab (Avastin) for Diabetic Retinopathy: The 2010 GLADAOF Lecture. J Ophthalmol. 2011;2011:584238. doi: 10.1155/2011/584238. Epub 2011 Mar 30. PMID 21584260
- [Background] Manzano RP, Peyman GA, Khan P, Kivilcim M. Testing intravitreal toxicity of bevacizumab (Avastin). Retina. 2006 Mar;26(3):257-61. doi: 10.1097/00006982-200603000-00001. PMID 16508423